CLINICAL TRIAL: NCT07049913
Title: GORE® TAG® Thoracic Branch Endoprosthesis Zone 2 Post-Market Surveillance in Japan
Brief Title: TBE Zone 2 PMS in Japan
Status: Recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 25-01
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Aneurysm Thoracic; Dissection of Aorta, Thoracic; Trauma
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TBE
  Interventions: Device: Gore® TAG® Thoracic Aortic Branch Stent Graft System

INTERVENTIONS:
Device: Gore® TAG® Thoracic Aortic Branch Stent Graft System — Patients who attempted implant of TBE in Zone 2 during the enrollment period of this surveillance.

SUMMARY:
The goal of this surveillance is to confirm the TBE device's safety and efficacy in patients treated with proximal landing in Zone 2 in the post-marketing period.

ELIGIBILITY:
Inclusion Criteria:

* Those who are suitable for use of TBE according to the Japan package insert.

[Reference: Purpose of Use or Effects of TBE at the time of launch] The GORE TAG Thoracic Branch Endoprosthesis is intended for use in patients with the following diseases with descending thoracic aortic lesions who fulfill anatomical requirements for treatment of such diseases while preserving blood flow to the left subclavian artery.

* Thoracic aortic aneurysm,
* Traumatic transection, and
* Complicated Stanford type B aortic dissection (including dissecting aortic aneurysm) who have not responded to medical therapy.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attempted implant of TBE in Zone 2 during the enrollment period of this surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2034-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Device Technical Success at the Initial Procedure | Initial procedure
  All of the following must be met.
  * Successful access and delivery
  * Patency of devices
  * The absence of unanticipated additional procedure related to the device, procedure, or withdrawal of the delivery system
Aortic Rupture of the Treatment Lesion | 60 Months
  Rupture in the treated segment of the vessel (e.g., aorta or branch) verified with direct observation or CT / CTA scan.
Lesion-related Mortality and All-cause Death | 60 Months
  Lesion-related Mortality definition
  Deaths that meet any of the following criteria:
  * All deaths within 30 days after the initial procedure during the initial hospitalization or secondary procedures resulting from the treated lesion or endovascular treatment (e.g., procedures for retrograde dissection, loss of patency, loss of device integrity, endoleak, migration, aortic dilation, aneurysm rupture)
  * All deaths related to the treated lesion or device (e.g., aneurysm rupture, retrograde dissection resulting in fatal cardiac tamponade) Not applicable if there is evidence to support no relationship to the lesion.
Disable Stroke | 60 Months
  Stroke is the acute onset of symptoms consistent with focal or multifocal central nervous system (CNS) injury caused by vascular blockage resulting in ischemia or vascular rupture resulting in hemorrhage, that:
  Persists for > 24 hours or until death
Serious Paraplegia | 60 Months
  Paraplegia secondary to spinal cord ischemia reported as a serious adverse event from sites.
Serious Paraparesis | 60 Months
  Paraparesis secondary to spinal cord ischemia reported as a serious adverse event from sites.
Renal Failure Requiring Dialysis | 60 Months
  Renal failure reported as a serious adverse event by sites and confirmed to require dialysis.
Additional Unanticipated Post-procedural Surgical or Interventional Procedure | 60 Months
  Additional unanticipated surgical procedure or endovascular procedure after the initial procedure.
  Anticipated or unanticipated status will be determined at the discretion of the investigator.
  Surgical procedures include conversion to thoracotomy, and endovascular procedures includes the placement of devices other than TBE.
  Endovascular procedures at the access site, lumbar drains for spinal cord ischemia, and procedures to address problems other than the treatment site (such as bare stent placement for intestinal ischemia due to dissection) do not apply.
Serious Device-related Ischemia | 60 Months
  Ischemia reported by sites as a serious adverse event determined to be related to the device.
Distal Device-related Thromboembolic Serious Adverse Event Requiring Intervention or Surgery | 60 Months
  Device-related ischemic adverse events reported by sites as serious adverse events that required bypass surgery, surgical procedures, or amputation, or that resulted in death.
Serious New Dissection | 60 Months
  New events of arterial dissection reported as serious adverse events by sites.
Serious Myocardial Infarction | 60 Months
  Myocardial infarction reported as a serious adverse event by the sites.
Serious Laryngeal or Phrenic Nerve Injury | 60 Months
  Nerve damage events reported by the sites as serious adverse events that required retreatment.
Serious Heart Failure/Hypotension | 60 Months
  Heart failure or hypotension reported as serious adverse events by the sites.
Aortic Enlargement in the Region Encompassed by the Initial Lesion | 60 Months
  An increase of 5 mm or more in arterial diameter at the affected area compared to images taken at the first follow-up after initial treatment.
Endoleak | 60 Months
  Serious adverse events reported or confirmed by imaging by the sites.
  The definitions of each type of endoleaks are as follows:
  * Type I endoleak is defined as a sealing failure at one of the attachment sites of the graft to the vessel wall. Arterial flow therefore leaks alongside the graft and into the perigraft space.
  * Type Ia: Proximal leak
  * Type Ib: Distal leak
  * Type Ic: Inadequate seal at distal landing zone for side branch component
  * Type II endoleak is defined as retrograde flow from branch arteries arising from the treated segment of the aorta.
  * Type III endoleak
  * Type IIIA endoleak : Attachment of aortic components (aortic-aortic).
  * Type IIIB endoleak : Fabric tear or disruption.
  * Type IIIC endoleak:: Attachment of aortic component-side-branch or side-branch-side-branch
  * Type IV endoleak is defined as flow through porous fabric.
  * Indeterminate : Endoleak detected with unknown source.
Loss of Device Integrity | 60 Months
  Defined as any of the following:
  * Wire fractures identified in the sealing row stents of the aortic component (AC), branch component (SB) or aortic extender (AE).
  * Stent kinking: Narrowing of the stent graft associated with demonstrable angulation in any of the stent components, with demonstrable flow
  * Disruption / tears in the graft component of the stent graft
  * Transient (compression) or permanent stent-graft collapse (invagination) following complete device deployment, resulting in an overall reduction in the aortic or branch vessel luminal diameter.
  * If the device loses function due to other malfunctions
Loss of Aortic or Aortic Branch Patency | 60 Months
  No flow or contrast detected through the implanted aortic or side branch devices or distal CTAG devices after the index endovascular procedure.
Migration | 60 Months
  Longitudinal movement of all or part of the device for a distance ≥10 mm, as confirmed by CT scan, relative to anatomical landmarks and device positioning at the first post-operative CT scan.
False Lumen Perfusion through the Primary Entry Tear (Dissection Patients only) | 60 Months
  Flow from a proximal aortic source through the primary intimal tear into the aortic false lumen (similar to a Type IA endoleak after treatment of aneurysms).
Extension of a Dissection (Proximally or Distally) (Dissection Patients only) | 60 Months
  Among the aortic dissections reported by sites as serious adverse events, those in which proximal or distal progression of the lesion from the initial procedure was confirmed on imaging.
False Lumen Status in Treated and Untreated Segments (Dissection Patients only) | 60 Months
  The thrombosis state of the false lumen at the treated and untreated segments at the initial procedure is confirmed using the following three stages.
  * Patent is defined as flow present throughout the aortic false lumen in the absence of evidence of thrombus.
  * Partially thrombosed false lumen is defined as clot within the aortic false lumen that has a residual patent flow channel.
  * Thrombosed false lumen is defined as complete thrombosis of the aortic false lumen.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Osaka Hospital, Osaka, Suita, Japan

IPD SHARING:
Plan to Share IPD: No